CLINICAL TRIAL: NCT04411446
Title: Randomized Controlled Trial of High Dose of Vitamin D as Compared With Placebo to Prevent Complications Among COVID-19 Patients
Brief Title: Cholecalciferol to Improve the Outcomes of COVID-19 Patients
Acronym: CARED
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Vitamin D Study Group (Network)
Collaborators: Agencia Nacional de Investigación y Desarrollo (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 001
Record Dates: First submitted 2020-05-26; First posted 2020-06-02 (Actual); Last update posted 2021-07-30 (Actual); Status verified 2021-03

CONDITIONS: COVID
Keywords: COVID; coronavirus; SARS-CoV-2; Vitamin D; Cholecalciferol; Respiratory insufficiency
MeSH Terms: conditions — Coronavirus Infections; Respiratory Insufficiency | interventions — Vitamin D; Cholecalciferol

STUDY DESIGN:
Intervention Model Description: Two parallel arms randomized controlled trial. A sequential design will be used with the first primary outcome being the primary outcome for the first step. This step will include 200 patients. After reach this point, a review of the primary outcome (change in respiratory SOFA) will be done. According to these results, the Executive committee will decide to proceed the second step of the study and include the remaining 1064 patients to evaluate the second primary outcome (need for high dose of oxygen supplementation or mechanical ventilation).
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The study will use a placebo identical to the active medication. The members of research team assessing the outcomes will not be aware of the treatment assignment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Vitamin D (Experimental): 5 capsules containing 100.000 UI of vitamin D each. The intervention will be 5 capsules given in one-time oral intake.
  Interventions: Drug: Vitamin D
- Placebo (Placebo Comparator): 5 capsules containing placebo. The intervention will be 5 capsules given in one-time oral intake.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Vitamin D — 5 capsules of 100.000 UI Vitamin D orally given all at once. One dose.
  Other Names: Cholecalciferol
  Arms: Vitamin D
Drug: Placebo — 5 capsules of containing placebo orally given all at once. One dose.
  Arms: Placebo

SUMMARY:
The recent inception of the coronavirus SARS-CoV-2, responsible for the coronavirus disease (COVID-19), has caused thousands of deaths globally. The most frequently reported complications among COVID-19 patients are from respiratory involvement.

Vitamin D has immunomodulatory effects that could protect against COVID-19 infection. Indeed, there is good evidence from randomized clinical trials suggesting that high doses of vitamin D administered during cold seasons prevent viral respiratory infections in at risk individual, and more recently, observational studies suggested that the mortality rate from COVID-19 is inversely correlated with levels of serum 25(OH)vitamin D.

The hypothesis of the study is that a high dose of vitamin D given orally to patients admitted to the hospital for COVID-19 will prevent the occurrence of respiratory deragement and other adverse clinical events.

To evaluate the aforementioned hypothesis, a randomized, controlled, double-blind, clinical trial comparing a 500.000 UI dose of vitamin D versus placebo among COVID-19 patients at moderate risk, requiring hospitalization but without requirements of critical care at admission was designed. The intervention will be one dose of 500.000 UI given orally or matching placebo.

The trial has a sequential design with two steps:

* The first step, projected to include 200 patients, will assess the effects of the intervention on the respiratory SOFA; and
* If there is a detectable effects, the second step, projected to include 1264 patients, will assess the effects on a combined event that includes need of high dose of oxygen or mechanical ventilation.

All study outcomes will be measured during the index hospitalization.

DETAILED DESCRIPTION:
See above.

ELIGIBILITY:
Inclusion Criteria:

* SARS-CoV-2 confirmed infection;
* Admission to a hospital;
* Expected hospitalization in the center for at least for 24 hs;
* Oxygen Saturation >90% breathing without oxygen supplement;
* Age at least 45 years or the presence of one of the followings risk factors:
* Hypertension;
* Diabetes (type I o II);
* At least moderate COPD or Asthma;
* Cardiovascular disease (history of myocardial infarction, coronary angioplasty, coronary artery bypass grafting or valve replacement surgery);
* Body Mass Index >=30;
* Signed Written consent.

Exclusion Criteria:

* <18 years old;
* Women in childbearing age;
* >= 72 hs since current admission;
* Requirement for high dose of oxygen (>5 liters/minute) or mechanical ventilation (non-invasive or invasive);
* History of Chronic kidney disease requiring hemodialysis or chronic liver failure;
* Inability for oral intake;
* Previous treatment with pharmacological vitamin D;
* History of:
* previous treatment with anticonvulsants;
* sarcoidosis;
* malabsorption syndrome;
* Known hypercalcemia.
* Life expectancy less than 6 months;
* Known allergy to the study medication;
* Any condition impeding to bring informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 218 (Actual)
Dates: Start 2020-08-11 (Actual); Primary Completion 2021-07-28 (Actual); Study Completion 2021-07-28 (Actual)

PRIMARY OUTCOMES:
Respiratory SOFA. | One week
  Is the respiratory component of the sequential organ failure assessment score (SOFA score). It is a 4 points scale, each point indicate a deeper respiratory impairment. The score is based on the relationship between the arterial pressure of oxygen (PaO2) and inspired fraction of oxygen (FiO2), as the ratio of both (PaFi). In the cases were arterial blood gas are not measured, the pulse oximetry will be used instead.
  The respiratory SOFA is as follows:
  * 1: PaO2/FiO2 >=300;
  * 2: PaO2/FiO2 >=200 and <300;
  * 3: PaO2/FiO2 >=100 and <200;
  * 4: PaO2/FiO2 <100.
  The minimum respiratory SOFA score will be record on daily basis during first week or to death or discharge, whichever occur first.
  This outcome is the primary outcome of the first study phase.
Need of a high dose of oxygen or mechanical ventilation. | 30 days
  The start of oxygen supplementation at FiO2 >40% or the initiation of invasive through orotracheal intubation) or non-invasive ventilation (Continuous positive airway pressure or Bilevel positive airway ventilation).
  This outcome will be recorded during hospitalization to 30 days, the death or discharge, whichever occur first.
  This is the primary outcome of the second study phase.

SECONDARY OUTCOMES:
Change in oxygen saturation. | One week
  Difference between the oxygen saturation at study entry and the lowest oxygen saturation measured during the first week, the death or discharge, whichever occur first.
  The oxygen saturation will be measured by pulse oximetry using commercially available devices.
Oxygen desaturation. | One week
  Oxygen saturation equal or less than 90% in any moment during the hospitalization. This outcome will be measured by pulse oximetry using commercially available devices.
  The outcome will be measured during the first week, the death or hospital discharge, whichever occur first.
Change in Quick SOFA score. | 30 days.
  The difference between the Quick SOFA score at study entry and the highest value recorded during the hospitalization.
  The outcome will be measured during the hospitalization until 30 days, the death or discharge whichever occur first.
Myocardial infarction. | 30 days
  Myocardial infarction is defined as suspicious symptoms with new Q waves in the EKG and enzymatic elevations compatible with the Fourth MI Definition.
  The outcome will be measured during the hospitalization until 30 days, the death or discharge whichever occur first.
Stroke. | 30 days
  Stroke is defined as a focal neurological loss lasting >24 hs as reported by treating physician.
  The outcome will be measured during the hospitalization until 30 days, the death or discharge whichever occur first.
Acute kidney injury. | 30 days
  Acute kidney injury is defined as an increase of at least 50% in serum creatinine levels (as compared with any previous value during the hospitalization).
  The outcome will be measured during the hospitalization until 30 days, the death or discharge whichever occur first.
Pulmonary thromboembolism. | 30 days
  Pulmonary thromboembolism is defined as the presence of suspicious symptoms (i.e. dyspnea) confirmed with objective evidence of a thrombus in the pulmonary tree by CT or MRI or Pulmonary Angiography.
  The outcome will be measured during the hospitalization until 30 days, the death or discharge whichever occur first.
Combined endpoint (stroke, myocardial infarction, acute kidney injury and pulmonary thromboembolism. | 30 days
  Combined outcome of the aforementioned events, Stroke is defined as a focal neurological loss lasting >24 hs as reported by treating physician.
  Myocardial infarction is defined as suspicious symptoms with new Q waves in the EKG and enzymatic elevations compatible with the Fourth MI Definition.
  Pulmonary thromboembolism is defined as the presence of suspicious symptoms (i.e. dyspnea) confirmed with objective evidence of a thrombus in the pulmonary tree by CT or MRI or Pulmonary Angiography.
  Acute kidney injury is defined as an increase of at least 50% in serum creatinine levels (as compared with any previous value during the hospitalization).
  The outcome will be measured during the hospitalization until 30 days, the death or discharge whichever occur first.
Admission to ICU. | 30 days
  Admission to Intensive Care Unit due to clinical deterioration as judged by the treating physician.
  The outcome will be measured during the hospitalization until 30 days, the death or discharge whichever occur first.
Invasive Mechanical Ventilation. | 30 days
  The start of mechanical ventilation invasive during the hospitalization until 30 days, the death or discharge whichever occur first.
Hospital Length of Stay. | 30 days.
  Total duration of initial hospital stay in days. The outcome will be measured during the hospitalization until 30 days, the death or discharge whichever occur first.
  In the cases with hospital stays longer than 30 days, it will considered as 30 days.
ICU length of stay. | 30 days
  Total duration of initial ICU stay in days. The outcome will be measured during the hospitalization until 30 days, the death or discharge whichever occur first.
  In the cases with ICU stays longer than 30 days, it will considered as 30 days.
Death | 30 days.
  Death of any cause during the hospitalization until 30 days or discharge whichever occur first.

CONTACTS AND LOCATIONS:
Overall Officials: Walter Manucha, PhD, Study Director — IMBECU, Univ Nac de Cuyo, Mendoza, Argentina; Carlos Tajer, MD, Principal Investigator — Hospital de Alta Complejidad El Cruce - Universidad Nacional Arturo Jauretche; Laura Antonietti, MD, Principal Investigator — Hospital de Alta Complejidad El Cruce - Universidad Nacional Arturo Jauretche; León Ferder, MD, Principal Investigator — Maimonides University; Felipe Inserra, MD, Principal Investigator — Universidad Maimónides - Hospital Universitario Austral; Javier Mariani, MD, Principal Investigator — Hospital de Alta Complejidad El Cruce - Universidad Nacional Arturo Jauretche
Locations (1):
- Hospital de Alta Complejidad en Red El Cruce, San Juan Bautista, Buenos Aires, Argentina

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Martin Gimenez VM, Inserra F, Tajer CD, Mariani J, Ferder L, Reiter RJ, Manucha W. Lungs as target of COVID-19 infection: Protective common molecular mechanisms of vitamin D and melatonin as a new potential synergistic treatment. Life Sci. 2020 Aug 1;254:117808. doi: 10.1016/j.lfs.2020.117808. Epub 2020 May 15. PMID 32422305
- [Derived] Mariani J, Antonietti L, Tajer C, Ferder L, Inserra F, Sanchez Cunto M, Brosio D, Ross F, Zylberman M, Lopez DE, Luna Hisano C, Maristany Batisda S, Pace G, Salvatore A, Hogrefe JF, Turela M, Gaido A, Rodera B, Banega E, Iglesias ME, Rzepeski M, Gomez Portillo JM, Bertelli M, Vilela A, Heffner L, Annetta VL, Moracho L, Carmona M, Melito G, Martinez MJ, Luna G, Vensentini N, Manucha W. High-dose vitamin D versus placebo to prevent complications in COVID-19 patients: Multicentre randomized controlled clinical trial. PLoS One. 2022 May 27;17(5):e0267918. doi: 10.1371/journal.pone.0267918. eCollection 2022. PMID 35622854
- [Derived] Mariani J, Tajer C, Antonietti L, Inserra F, Ferder L, Manucha W. High-dose vitamin D versus placebo to prevent complications in COVID-19 patients: A structured summary of a study protocol for a randomised controlled trial (CARED-TRIAL). Trials. 2021 Feb 1;22(1):111. doi: 10.1186/s13063-021-05073-3. PMID 33522946